CLINICAL TRIAL: NCT02043158
Title: Biobehavioral and Sociodemographic Characteristics of Long Term Survivors of Ovarian Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2013-0626; 1234 (Other: Department of Defense); NCI-2021-10800 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Short term survivors; Long term survivors; Biobehavioral characteristics; Sociodemographic characteristics; Questionnaire; Survey; Interview
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian Cancer Survivors: Short-term and long-term ovarian cancer survivors
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire completion asking questions about quality of life, mood, social support, stress, diet, lifestyle, and demographic information. Questionnaire should take about 60-90 minutes to complete.
  Other Names: Survey
Behavioral: Interview — Interview asking questions about the amount of stress participant may be having or have had in the past. It should take about 25-30 minutes to complete the interview.

SUMMARY:
The goal of this research study is to learn about diet and exercise habits, emotions, and social support in the lives of women with ovarian cancer.

DETAILED DESCRIPTION:
Study Participation:

If you agree to take part in this study, you will fill out a questionnaire, complete an interview, and information will be collected from your medical record.

For the questionnaire, you will answer questions about your quality of life, mood, social support, stress, diet, lifestyle, and demographic information (such as your age and race). The questionnaire should take about 60-90 minutes to complete. If you prefer to fill out the questionnaire online, 3 separate emails will be sent to your email address. Each email will contain a separate link (the first link will be sent from MD Anderson, the second from University of Arizona for the diet questions, and the third from the University of California Los Angeles [UCLA] for the stress questions).

You will also be asked to measure your waist and your hip with a measuring tape and to record the measurements on the questionnaire.

If you prefer to fill out the questionnaire by paper format, you should mail it back to the research staff. However, the stress questions will need to done by phone. A trained interviewer will ask you questions about the amount of stress you may be having or have had in the past. It should take about 25-30 minutes to complete the interview.

If you are a long-term survivor, you will have an interview by phone that will ask for your opinions about the factors that may have contributed to your survival. This interview will take about 45 minutes to an hour and will be audio-recorded. Your name and identifying information will not be recorded.

Information collected from your medical record will include the status of the disease, if the disease has gotten worse, any treatments you have received, and any side effects you may have had. This information will help researchers learn how specific treatments may affect patients.

If you are already enrolled in a protocol in which you will be having tumor tissue collected for future analysis, the information gathered in those studies will be used together with the data collected for this study to learn if behavioral factors relate to your tumor tissue test results.

Length of Study:

Your study participation will be over after completing the questionnaire and interview.

Other Information:

Before any information is recorded, you will be asked for your permission.

The tape recording will be done by members of the study staff. Your audiotape will be given a code number. No identifying information (such as your name and medical record number) will be recorded on the audiotape.

This is an investigational study.

Up to 240 participants will be enrolled in this multicenter study. Up to 120 will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. For the long-term survivor group: alive for at least seven years post-diagnosis.
2. At least 18 years of age.
3. Can speak and read English.
4. diagnosed with stage III-IV ovarian, peritoneal or fallopian tube cancer

Exclusion Criteria:

1. Are in hospice or about to be referred to hospice within the next 3-6 weeks.
2. Are not oriented to time, person, or place.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Long term and short term ovarian cancer survivors at the University of Texas MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2014-01-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Biobehavioral Information Collection in Ovarian Cancer Survivors | 1 day
  Biobehavioral information collected regarding social support, depressed mood, life stress, quality of life, meaning in life, socioeconomic and relationship status, and lifestyle factors such as exercise and diet, which have been linked with cancer progression and/or survival in cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H. Shinn, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Cedars Sinai, West Hollywood, California
  - University of Iowa, Iowa City, Iowa
  - Memorial Sloan Kettering, New York, New York
  - University of Oklahoma, Norman, Oklahoma
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org